CLINICAL TRIAL: NCT00380952
Title: MAST Study Protocol
Brief Title: Intraoperative Use of the BP Device for Detecting Positive Margins During Lumpectomy Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dune Medical Devices (Industry)
Responsible Party: Orit Yarden, Medical VP
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-02-001
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Breast Cancer
Keywords: IDC; DCIS; ILC
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Dune Device

SUMMARY:
This protocol was designed for testing the intraoperative use of the Dune device. This multicenter study will take place in Israel at 12 sites.

DETAILED DESCRIPTION:
Use of the device will take place during a partial mastectomy procedure (lumpectomy).The patient will be randomized to enter the device or control arm.

ELIGIBILITY:
Inclusion criteria

1. Women diagnosed with carcinoma of the breast
2. Undergoing lumpectomy (local wide excision) procedure.
3. Over 18 years of age
4. Signed ICF

Exclusion criteria

1. Neoadjuvant systemic therapy
2. Previous radiation in the operated breast
3. Prior surgical procedure in the same quadrant
4. Implants in the operated breast
5. Pregnancy
6. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-11; Primary Completion 2007-10 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Hershko, Dr., Principal Investigator — Rambam MC; Rona Spector, Dr., Principal Investigator — Rabin MC; Eran Sharon, Principal Investigator — Rabin MC; Zvi Kaufman, Dr., Principal Investigator — Meir MC; Tal Kopelman, Dr., Principal Investigator — Bnei Zion Mc; Yuri Berlin, Dr., Principal Investigator — HaEmek MC; Moshe Papa, Prof., Principal Investigator — Sheba Mc; Tanir Allweis, Dr., Principal Investigator — Haddasah Medical Organization; Shlomo Schneebaum, Prof., Principal Investigator — Souraski MC; Moshe Carmon, Dr., Principal Investigator — Shaare Zedek MC; Amram Adari, Dr., Principal Investigator — Ziv Mc; Moshe Zilberman, Dr., Principal Investigator — Poria MC
Locations (9):
- Israel (9):
  - HaEmek Mc, Afula
  - Rambam MC, Haifa
  - Haddasah Medical Organization, Jerusalem
  - Shaare Zedek, Jerusalem
  - Meir MC, Kfar Saba
  - Rabin MC, Petah Tikva
  - Rivka Ziv MC, Safed
  - Souraski MC, Tel Aviv
  - Poria MC, Tiberias

REFERENCES:
- See also: Official company site — http://www.dunemedical.com